CLINICAL TRIAL: NCT06957457
Title: The Effect of Music Accompanied Aerobic Exercise on Pain, Quality of Life and Well-Being in Patients With Fibromyalgia Syndrome
Brief Title: The Effect of Music Accompanied Aerobic Exercise
Acronym: Music
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Berna Dincer, Nursing Associate Professor, Istanbul Medeniyet University
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IstanbulMU
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Fibromyalgia; Fibromyalgia (FM); Syndrome Pain; Exercise
Keywords: fibromyalgia; syndrome; exercise
MeSH Terms: conditions — Fibromyalgia; Somatoform Disorders; Motor Activity; Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Assuming a power of 80% and an α risk of. 05, a sample size of 75 was determined to be appropriate. Considering the possibility of missing data, the study initially included 80 participants in both the experimental and control groups. A computer-based random number generator was used for group assignment, and allocation concealment was ensured by using sealed envelopes containing random numbers opened by a separate researcher. The study was completed with 40 participants in the experimental group and 40 in the control group, due to some participants withdrawing.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: exercise (Experimental): Do Exercise
  Interventions: Behavioral: Exercise
- Control (Active Comparator): do nothing
  Interventions: Behavioral: Control (Standard treatment)

INTERVENTIONS:
Behavioral: Exercise — The exercise program lasts 32 minutes in total. The first 6 (six) minutes of this program consists of warm-up exercises. Active exercise time is 21 (twenty-one) minutes. Relaxation exercises consist of 5 (five) minutes of relaxation exercises. exercise was accompanied by music. it consists of warm-up exercise and relaxation sections.
  Arms: Experimental: exercise
Behavioral: Control (Standard treatment) — do nothing
  Arms: Control

SUMMARY:
Objective: The aim of this study, which was planned as a single-blind randomized controlled design, was to investigate whether aerobic exercise accompanied by music has positive effects on pain, quality of life and well-being in patients with fibromyalgia syndrome.

Materials and Methods: The study sample consisted of 80 patients diagnosed with fibromyalgia syndrome The patients were randomly assigned to either the experimental (n=40) or control group (n=40) using a computer-based randomization method. Data collection tools included the Personal Information Form , Fibromyalgia Impact Questionnaire Scale , State Anxiety Scale (STAI-I/STAI II) , Psychological Well-Being Scale

DETAILED DESCRIPTION:
Objective: The aim of this study, which was planned as a single-blind randomized controlled design, was to investigate whether aerobic exercise accompanied by music has positive effects on pain, quality of life and well-being in patients with fibromyalgia syndrome.

Materials and Methods: The study sample consisted of 80 patients diagnosed with fibromyalgia syndrome The patients were randomly assigned to either the experimental (n=40) or control group (n=40) using a computer-based randomization method. Data collection tools included the Personal Information Form , Fibromyalgia Impact Questionnaire Scale , State Anxiety Scale (STAI-I/STAI II) , Psychological Well-Being Scale

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with fibromyalgia according to the 2016 American College of Rheumatology criteria in the Physical Therapy and Rehabilitation unit of the University of Health Sciences Kanuni Sultan Süleyman Training and Research Hospital,
* Being between the ages of 18 and 65,
* Volunteering to participate in the study.
* Having no problem with perception
* Being diagnosed with fibromyalgia at least 6 (six) months ago.
* Not using any alternative treatment method (acupuncture, mud, etc.).

Exclusion Criteria:

* Cardiovascular, respiratory, metabolic and rheumatic diseases that may limit exercise;
* Diseases associated with autonomic dysfunction such as arterial hypertension, diabetes and coronary insufficiency;
* Having exercised in the last 3 months,
* Having a disease that causes problems in understanding the questionnaires
* Pregnancy or breastfeeding.
* History of surgery in the last four months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-11-23 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire Scale | up to 4 weeks
  The first item in the questionnaire includes a scale of 0-3 (0: always 1: most of the time 2: sometimes 3: never) for 11 activities of daily living such as shopping, laundry, cooking, making beds, washing dishes by hand, vacuuming carpets, walking a few blocks, visiting friends/relatives, gardening, driving, and climbing stairs. The second and third items ask about well-being and the number of days of problems due to illness. The next seven items assess the patients' ability to work, pain intensity, fatigue, stiffness, good sleep, anxiety and depression during the previous week using VAS. The maximum total score is 100. High scores indicate low functionality of the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No